CLINICAL TRIAL: NCT05859100
Title: Can Protein Intake be Increased Using Whole Foods Post-treatment in Cancer Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Egg Farmers of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-22-0348
Record Dates: First submitted 2023-04-13; First posted 2023-05-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Other Malnutrition
Keywords: Cancer; Nutrition; Protein; post-chemotherapy; Recovery; food-related quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two parallel arms (i.e., egg intervention arm and no intervention arm) for the first 4 weeks. Starting from week 5, the participants in the egg intervention arm will continue with the intervention till week 8 and the participants in the control arm will crossover to the intervention arm for weeks 5 to 8.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Experimental): Participants are expected to begin intervention immediately after the completion of treatment for a period of 8 weeks.
  Interventions: Other: ≥ 2 eggs in addition to usual diet for 8 weeks
- Delayed Intervention (Other): Participants are expected to begin intervention 4 weeks after the completion of the treatment, for a period of 4 weeks (weeks 5-8).
  Interventions: Other: ≥ 2 eggs in addition to usual diet for 4 weeks

INTERVENTIONS:
Other: ≥ 2 eggs in addition to usual diet for 8 weeks — Participants are expected to consume≥ 2 eggs per day in addition to usual diet for 8 weeks in early intervention arm, beginning immediately post-treatment.
  Arms: Early Intervention
Other: ≥ 2 eggs in addition to usual diet for 4 weeks — Participants are expected to continue intake of regular diet beginning immediately at post-treatment recovery for a duration of 4 weeks, then crossover to nutritional intervention arm from weeks 5 to 8 of post-treatment recovery for a duration of 4 weeks.
  Arms: Delayed Intervention

SUMMARY:
Cancer and its treatments often result in severe toxicities and side effects that, over the course of treatment, results in weight loss and depletion of key nutrients. Loss of muscle mass and strength during cancer treatment is a critical problem because it negatively affects patient response and tolerance to therapy and post-treatment recovery. To restore the nutritional status, it is imperative to stimulate muscle protein anabolism. Eggs are high quality protein source, popular and well tolerated by cancer patients. Therefore, the objective of this study is to determine whether a nutritional intervention of ≥2 eggs can aid in restoring nutritional status and improving immune function and quality of life of cancer patients' post-treatment. It is an 8- week randomised clinical trial with parallel arm assignment. Half of the participants will receive the nutritional intervention (Early Intervention) and the other half will be on standard of care or usual diet for first 4 weeks. Starting from week 5, all participants will receive the nutrition intervention till week 8 (Delayed Intervention). Dietary intake (foods and nutrients), cumulative protein intake (g protein/kg body weight), immunological measures, physical performance and quality of life has been planned to be assessed over time and between groups to evaluate the feasibility of an egg intervention in meeting recommended protein intakes for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.
* ≥18 years of age
* Histopathologically confirmed cancer with receipt of a platinum chemotherapy during treatment; active treatment has concluded.
* Capable of volitional oral semi-solid intake at baseline; able to maintain oral intake over the trial.

Exclusion Criteria:

* Fed by nasogastric tube, gastrostomy, or total parenteral nutrition
* Cancer of the brain, Cancer of the regions which impact an individual's ability to consume food.
* A known hypersensitivity / allergy to eggs.
* Enrolment in any other clinical protocol or investigational study that may interfere with study procedures.
* Poorly controlled chronic illnesses or other inflammatory diseases (e.g. Chronic Obstructive Pulmonary Disease(COPD), uncontrolled non-insulin dependent diabetes, rheumatoid arthritis).
* In a clinician opinion, patients who have medical conditions that could interfere with nutrient metabolism or absorption (e.g., short bowel syndrome, Crohn's disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Difference in mean cumulative protein intake between the two groups at 8 weeks. | From baseline at 8 weeks
  Mean cumulative protein intake will be arrived at by normalizing protein intake in kilocalories by body weight in kilograms
Difference in mean cumulative protein intake within a group at 8 weeks for each group. | From baseline at 8 weeks
  Mean cumulative protein intake will be arrived at by normalizing protein intake in kilocalories by body weight in kilograms

SECONDARY OUTCOMES:
Change in Energy Intake | From baseline at 8 weeks
  Energy intake can be described as energy intake in kilocalories normalized by body weight in kilograms.
Change in Body weight | From baseline at 8 weeks
  in kilograms
Change in Quality of Life | From baseline at 8 weeks
  Research and Development(RAND) Short Form 36-Item Health Survey 1.0 Minimum to Maximum score= 0 to 100 High Score indicates more favorable outcome.
Change in Nutritional status and Symptom severity. | From baseline at 8 weeks
  Patient generated-subjective global assessment (PG-SGA), 0-9 point score, higher the score more severe the malnourishment.
  Edmonton Symptom Assessment Scale- Revised (ESAS-r, 0 to 10 Visual analog scale, higher the number more severe the symptom)
Change in Quality of Life related to malnutrition | From baseline at 8 weeks
  Functional assessment of Anorexia-Cachexia Therapy 5 question Anorexia/ Cachexia subscale (FAACT A/C Subscale, Score Range= 0 to 20, Higher the score better the quality of life)
Change in Physical performance | From baseline at 8 weeks
  Short physical performance battery (SPPB, Score range= 0 to 12, higher the score better the performance)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Mazurak, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No